CLINICAL TRIAL: NCT02244541
Title: Phase 2a Study of ANAVEX2-73 Adaptive-Trial-Design With Repeated Doses, MTD Finding, Pharmacodynamic and Bioavailability Evaluation in Patients With Mild to Moderate Alzheimer's Disease With a 12-Month Open Label Follow-Up Period
Brief Title: Phase 2a Dose Finding, PK/PD and 12 Month Exploratory Efficacy Study of ANAVEX2-73 in Patients With Alzheimer's Disease
Acronym: ANAVEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANAVEX2-73-002
Record Dates: First submitted 2014-08-31; First posted 2014-09-19 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tetrahydro-N, N-dimethyl-2,2-diphenyl-3-furanmethanamine hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Anavex2-73 oral then the Anavex2-73 intravenous formulation (Experimental): Participants first receive Anavex2-73 hard gelatin capsule each morning with a light breakfast for 11 days. After a washout period of 11 days they then receive the Anavex2-73 intravenous formulation each morning with a light breakfast for 11 days.
  Interventions: Drug: ANAVEX2-73 Oral; Drug: ANAVEX2-73 Intravenous
- Anavex2-73 intravenous then the Anavex2-73 oral formulation (Experimental): Participants first receive Anavex2-73 intravenous formulation each morning with a light breakfast for 11 days. After a washout period of 11 days then they receive the Anavex2-73 hard gelatin capsule each morning with a light breakfast for 11 days.
  Interventions: Drug: ANAVEX2-73 Oral; Drug: ANAVEX2-73 Intravenous
- Anavex2-73 30 mg oral formulation (Experimental): Participants will receive the 30 mg Anavex2-73 hard gelatin capsule orally once daily for 52 weeks.
  Interventions: Drug: ANAVEX2-73 Oral
- Anavex2-73 50 mg oral formulation (Experimental): Participants will receive the 50 mg Anavex2-73 hard gelatin capsule orally once daily for 52 weeks.
  Interventions: Drug: ANAVEX2-73 Oral

INTERVENTIONS:
Drug: ANAVEX2-73 Oral
  Arms: Anavex2-73 intravenous then the Anavex2-73 oral formulation; Anavex2-73 oral then the Anavex2-73 intravenous formulation
Drug: ANAVEX2-73 Intravenous
  Arms: Anavex2-73 intravenous then the Anavex2-73 oral formulation; Anavex2-73 oral then the Anavex2-73 intravenous formulation
Drug: ANAVEX2-73 Oral — 30 mg hard gelatin capsule
  Arms: Anavex2-73 30 mg oral formulation
Drug: ANAVEX2-73 Oral — 50 mg hard gelatin capsule
  Arms: Anavex2-73 50 mg oral formulation

SUMMARY:
The primary objective of this Phase 2a study is to evaluate the maximal tolerated dose of ANAVEX2-73 in patients with AD in a repeated-dose administration scheme, with the secondary objectives being to explore the relationship between dosing regimen and pharmacodynamics efficacy outcomes and to evaluate the bioavailability of the oral form used and to explore the relationship of ANAVEX2-73 as add-on therapy to AD standard of care.

DETAILED DESCRIPTION:
This is a Phase 2a study consisting of two parts, PART A and PART B. The first part (PART A) is a simple randomised, open-label, 2-period, cross-over, adaptive design study lasting for each participant up to 36 days.

The second part (PART B) is an open-label extension for an additional period of 52 weeks, so as to establish a longer drug effect for the participants who wish to continue on oral daily dose.

The complete timeline of the study includes the screening assessments within 28 days prior to simple randomisation and initiation of the study. The first administration of study medication will occur after all baseline and screening procedures have been passed (baseline is defined as pre-dosing period timeframe day -28 to day -1). No study procedures will be undertaken until a current informed consent form has been signed by each participant or their respective carer or responsible person.

The design of the first part (PART A) of the study involves two periods, two administration routes and two dose levels: In one period the intravenous (iv) form will be given and in the other period the oral dose will be given. The first period will involve 12 administrations (either oral or iv) and the second period will involve 11 administrations (either oral or iv).

The very first administration in the first period is intended as a full pharmacokinetic (PK) screen over the first 48 hours (Day 1 to Day 3). After that, 11 daily administrations complete the first period (Day 3 to Day 13). After a wash-out period of 11 days, the second period of the study starts, involving again 11 daily administrations. Therefore, the first part (PART A) of the study is scheduled to be completed in 36 days.

The study design asks for 32 participants, 16 males and 16 female participants. All participants have the option to go on to the second part (PART B) of the study, the extended open-label study exploring the cognitive effect of the drug for another 52 weeks where the oral form will be exclusively administered.

Safety and tolerability will be constantly assessed throughout the study, starting from the first dose of study medication.

ELIGIBILITY:
Main Inclusion Criteria:

1. Diagnosis of Probable AD in accordance with NINCDS-ADRDA criteria.
2. A brain CT or MRI scan performed within last 12 months from day of screening consistent with the clinical diagnosis of probable AD.
3. Age from 55 to 85 years inclusive.
4. MMSE score of 16-28 inclusive.
5. Rosen Modified Hachinski Ischemic score <=4.
6. Community dwelling with caregiver who has regular contact with the subject for at least 10 hours per week and is able to oversee the patient's compliance with study medication and participate in the patient's clinical assessment and is capable of accompanying the participant on all clinic visits.
7. Fluency in English.
8. Be able to read, write, speak clearly for the cognitive tests, with eyesight and hearing sufficient to enable completion of the cognitive tests.
9. Receiving stable doses of medications for the treatment of non-excluded medical conditions for at least 30 days prior to screening.

Main Exclusion Criteria:

1. Dementia other than AD such as AIDS, CJD, LBD, CVD, Progressive Supranuclear Palsy, Multiple cerebral infarcts, or normal pressure hydrocephalus.
2. Other neurodegenerative diseases, including Parkinson's disease and Huntington's disease, or cerebral tumour.
3. Current presence of a clinically significant major psychiatric disorder according to the criteria of the DSM-IV, or symptom that could affect the participant's ability to complete the study). HAM-D score >12.
4. Current clinically significant systemic illness that is likely to result in deterioration of the patient's condition or affect the patient's safety during the study.
5. Any other criteria which in the opinion of the Investigator causes the participant not to qualify for the study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
To determine maximum tolerated dose of Anavex2-73. | 36 Days

SECONDARY OUTCOMES:
PK sampling- blood test results | First part (PART A), first period (hours): 1, 48, 264; second period (hours): 1, 72, 264; extension period (PART B): Week 1, 12 and 26.
Mini-mental state examination score (MMSE) | Baseline, and during the extension period at Week 1, 12, 26, 36, 48, and 52
Score from ADCS-ADL (Alzheimer's Disease Co-operative Study - Activities of Daily Living Inventory) | Baseline, and during the extension period at Week 1, 12, 26, 36, 48, and 52
Cogstate Brief Battery (CBB) Score and International Shopping List Task (ISLT) Score | At baseline, Day 1, 2, 6, 9, 12 of Period 1 and Day 1, 2, 6, 9, 12 of Period 2 and during the extension period at Week 12, 36, 48, and 52.
Electroencephalographic activity, including event-related potentials (EEG/ERP) | baseline, Day 1, 5, 11 of Period 1 and Day 1, 5, 11 of Period 2 and, Week 12, 36, 48, and 52 of the extension period
Hamilton Psychiatric Rating Scale for Depression (HAM-D) Score | Baseline at Period 1
Rosen Modified Hachinski Ischemic Score (RM/HIS10) | Baseline at period 1

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Macfarlane, Principal Investigator — Caulfield Hospital
Locations (5):
- Australia (5):
  - Melbourne Health - The Royal Melbourne Hospital, Melbourne, Victoria
  - Austin Health - Heidelberg Repatriation Hospital, Melbourne, Victoria
  - Caulfield Hospital, Melbourne, Victoria
  - Nucleus Network- Centre for Clinical Studies, Melbourne, Victoria
  - St. Vincent's Hospital, Melbourne, Victoria